CLINICAL TRIAL: NCT05746936
Title: Can Robotic Gastric Bypass be Considered a Valid Alternative to Laparoscopy: Our Early Experience
Brief Title: Robotic Versus Laparoscopic Roux En-y Gastric Bypass
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Principal Investigator, University of Foggia
Other Study IDs: 7
Record Dates: First submitted 2023-02-02; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Roux-en-y Anastomosis Site; Obesity, Morbid; Bypass Complication; Anastomosis; Complications; Surgery-Complications
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients underwent laparoscopic gastric bypass
  Interventions: Procedure: Roux en-Y gastric bypass
- obese patients underwent robotic gastric bypass
  Interventions: Procedure: Roux en-Y gastric bypass

INTERVENTIONS:
Procedure: Roux en-Y gastric bypass — gastric bypass with jejuna-jenual anastomosis and gusto-jejunal anastomosis

SUMMARY:
This study retrospectively identified 33 consecutive obese patients who underwent either laparoscopic or robotic gastric bypass procedures over a 2-year period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥35-39 kg/m2 with one obesity- associated co-morbidity
* BMI≥40kg/m2, age ≥ 18 years.

Exclusion Criteria:

* Re-do surgery procedures

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Body mass index (BMI) ≥35-39 kg/m2 with one obesity- associated co-morbidity or BMI≥40kg/m2, age ≥ 18 years. Before surgery, patients underwent a standardized psychological and physical evaluation which includes blood chemistry tests, chest x-rays, electrocardiogram and cardiological examinations, nutritional evaluation, esophagogastroduodenoscopy, spirometry and psychiatric evaluation .
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
differences between the robotic and laparoscopic gastric bypass | two years period
  incidence of mortality and morbidity (percentage)
differences between the robotic and laparoscopic gastric bypass | two years period
  BMI ( kg/m2)
differences between the robotic and laparoscopic gastric bypass | two years period
  age (years)
differences between the robotic and laparoscopic gastric bypass | two years period
  weight (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavone G, Pacilli M, Gerundo A, Quazzico A, Ambrosi A, Tartaglia N. Can robotic gastric bypass be considered a valid alternative to laparoscopy? Our early experience and literature review. Front Surg. 2024 Feb 5;11:1303351. doi: 10.3389/fsurg.2024.1303351. eCollection 2024. PMID 38375411

DOCUMENTS (1):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT05746936/Prot_000.pdf